CLINICAL TRIAL: NCT04695457
Title: Correlation Between the Incidence of COVID-19 in Nursing-homes and the Profile of Nursing Homes in the French Alps
Acronym: PROCOPAD
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Annecy Genevois (Other)
Responsible Party: Sponsor
Other Study IDs: 20-13
Record Dates: First submitted 2020-12-08; First posted 2021-01-05 (Actual); Last update posted 2021-01-05 (Actual); Status verified 2021-01

CONDITIONS: Covid19; Nursing Home
Keywords: covid19; nursing home
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Since the beginning of the COVID-19 outbreak in France, nursing homes (NH) have been heavily affected. In this study, the investigators want to evaluate the factors associated with the occurrence of COVID-19 epidemic clusters within the nursing homes in the French Alps

DETAILED DESCRIPTION:
In France, between 1st of March and 29th of June 2020, the situation of NH was critical, with a total of 5,203 outbreaks (≥ 1case), of which 651 (13%) occurred in the Auvergne-Rhône-Alpes (ARA) area. In the ARA area, 3,885 residents of NH were confirmed cases (positiveness of the polymerase chain reaction (PCR) or of the serology testing), of which 1,772 (46%) subsequently died. To manage this crisis, the French government decided to first, ban the visits to residents and to reinforce hygiene measures targeting care workers, and secondly, of a national lock down. In the same time, shortage of personal protective equipment (PPE) had happened worldwide.

In this context, one can hypothesize that the occurrence of outbreaks and its spread among the residents of NH would have been initiated by the staff members. Nonetheless, the implementation of local actions might have been efficient to mitigate the epidemic, while on the other hand, shortage of PPE might have worsen the epidemic.

Therefore the investigators aimed to investigate the relationship between the occurrence of outbreak in residents and in staff members of nursing home, as well as the factors influencing this relationship, using data from a multicentric cross-sectional survey conducted in the French Alps, a part of ARA area.

ELIGIBILITY:
Inclusion Criteria:

* Hospital based NH in the French Alps
* Non Hospital based NH in the French Alps
* Study participation agreement from the NH's managers

Exclusion Criteria:

* Refusal of the NH's managers to participate

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: NH which are part of the French Alps in the ARA area.
  The questionnaire was made available on the internet 24 h/day, 7 days/week using the dedicated link sent to each NH through email by the research team on 15th of July. NH's managers had to respond to the survey.
Sampling Method: Probability Sample
Enrollment: 74 (Actual)
Dates: Start 2020-07-15 (Actual); Primary Completion 2020-11-16 (Actual); Study Completion 2020-11-16 (Actual)

PRIMARY OUTCOMES:
Identification of factors associated with the occurrence of COVID-19 outbreak in French Alps' nursing homes | day 1
  Establish the factors associated with the occurrence of clustered cases by comparing the structural and organizational characteristics of NHs having experienced grouped cases, that is to say having presented at least 3 cases of COVID-19 between March 01 and May 31, 2020 compared to NHs having no clustered cases of COVID-19 during this same period.
  Evaluation, using a regression model, on aggregated data, of the associations (univariate, multivariate) between the occurrence of grouped cases and the following criteria:
  * Type of NH (public or private);
  * The average degree of dependency and of morbidity of the residents (Gir Moyen Pondéré (GMP) and Pathos Moyen pondéré (PMP)) scales.
  * Number of residents in the NH;
  * Human resources used during the epidemic:
  * Operational management of the crisis: date of visit ban, face mask's wearing condition for the personnel
  Associations measured using "odds ratios" and their 95% confidence interval (95% CI).

CONTACTS AND LOCATIONS:
Locations (1):
- Ch Annecy Genevois, Pringy, France